CLINICAL TRIAL: NCT01809509
Title: A Prestudy of Impact of Cytokines and Gene Expression on Outcome of IVF
Brief Title: Pilot Study on Molecular Quantitation and Sequencing of Endometrial Cytokines Gene Expression and Their Effect on the Outcome of In-vitro Fertilization (IVF) Cycle
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Nooh Riad Ali, assistant professor Cairo university, Cairo University
Other Study IDs: FDAAA
Record Dates: First submitted 2013-03-09; First posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Endometrial Receptivity and Success Rate of IVF
Keywords: CYTOKINES , IL11 IL6 IMLANTATION RATE IVF.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endometrial biopsy

SUMMARY:
Pilot study on molecular quantitation and sequencing of endometrial cytokines gene expression and their effect on the outcome of in-vitro fertilization (IVF) Cycle

DETAILED DESCRIPTION:
The study will be performed

in the Cairo IVE Unit; Faculty of medicine Cairo University on 15 cases. Inclusion criteria: age 23 -35, FSH less than 10 no previous uterine operations, no history of poor response in previous IVF no sever male factor no endometriosis and uterine factor are excluded . no diabetes mellitus and antral follicle count (AFC) > 5 undergoing IVF using standard long protocol.

All patients will give their informed consent to participate in the study. Endometrial tissue samples will be taken on the day of oocyte retrieval using soft suction plastic catheter. The menstrual blood of 10 women with regular menstrual cycles and with no apparent endometrial dysfunction was taken as control samples. The study protocol and informed consents were approved by the Human Ethics Committee of IVF department .of Kasar Ini hospital

Total RNA isolation: Endometrial biopsies and menstrual control blood will be lysed by RLT buffer (QIAGEN, Germantown, MD). The lysates further prepared for total RNA extraction using the RNeasy mini kit (QIAGEN, Germantown, MD) according to the manufacturer's instructions. The RNA extract stored at -80ºC until future use. RNA purity, yield, and concentration will be determined through dual spectrophotometry (Beckman, USA), and 1μg of RNA run on a 1% agarose gel (Roche, Castle Hill, Australia) to ensure integrity of the RNA. Quantitative RT-PCR (qRT-PCR): Reverse transcriptase (RT) reaction mixture using High Capacity Reverse Transcriptase kit (Applied Biosystems, USA) containing: 1 μg total RNA from each sample for cDNA synthesis, 0.5 μg random primer, 5×RT buffer, 2.5 mmol/L dNTP, 20 U RNase inhibitor and 200 U MMLV reverse transcriptase in a total volume of 25 μl was incubated at 37ºC for 60 minutes, then heated to 95 ºC for 5 minutes to inactivate MMLV. RT will be followed by qPCR, 50 ng of cDNA were added to 5 X Fast-Start SYBR green master mix with Rox (Roche Diagnostics, Indianapolis, IN) and 200 ng of primer mix (Sigma). The reaction will be carried out in micro optical plates (Applied Biosystems) and analyzed using StepOne real-time 203 PCR system (Applied Biosystems). The PCR running method was as follows: 10 minutes at 950C for enzyme activation followed by 40 cycles of 15 seconds at 950C, 20 seconds at 550C and 30 second at 720C for the amplification step. The primers used in the qRT-PCR evaluation specific for target genes (table 1). Relative mRNA expression will be calculated by the comparative cycle threshold method . as outlined in the manufacturer's user manual with GAPDH house-keeping gene. The fluorescence was plotted versus PCR cycle number for reaction and each sample indicated. Serum hormonal levels assay: FSH, LH and E2 were estimated by ELISA according to instructions of manufacturers. DNA purification and sequencing analysis: IL-11 and LIF genes analyzed by direct sequencing of the PCR products using SEQr kit. (Applied Biosystems), according to manufacturer's protocol. PCR products will be purified using the QIAquick Gel Extraction Kit (QIAGEN). The relevant purified DNA samples of all the cases and controls will be amplified and sequenced using automated sequencing with the aid of a Big Dye Terminator Sequencing Kit (PE/Applied Biosystems, Foster City, CA). The samples will be run in an automated sequencer ABI Prism 310 Avant (PE/Applied Biosystems).. All samples will be sequenced twice to ensure the results.

Statistical analysis: Data will be statistically described in terms of mean standard deviation , median and range. Comparison between women who could achieve pregnancy and those who didn't was done using Mann Whitney U test for independent samples. Correlation between various variables was done using Spearman rank correlation equation for non-normal variables.

ELIGIBILITY:
Inclusion Criteria:

- FSH LESS THAN 10 ,

Exclusion Criteria:

NO SEVER MALE FACTOR no endometriosis , DM or previous uterine surgery .

Ages: 23 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: those under going IVF using standard protocol
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
relation between IL11 AND IL6 PRESENCE AND GENE EXPRESSION AND SUCCESS OF IVF | one year

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Olfat Nooh Riad Ali, Cairo
  - IVF centre, Cairo